CLINICAL TRIAL: NCT04854902
Title: The Effects of Cyanoacrylate on Self-reported Outcomes and Healing Following Free Gingival Graft Surgery
Brief Title: Cyanoacrylate Use in Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Mustafa YILMAZ, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAFGG
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession | interventions — Cyanoacrylates; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyanoacrylate (Experimental): The graft is stabilized and the donor site is coated with cyanoacrylate.
  Interventions: Procedure: Free gingival graft; Procedure: Cyanoacrylate
- Suture (Active Comparator): 6/0 polyvinylidene fluoride sutures are used for stabilization, while the donor site is left untreated.
  Interventions: Procedure: Free gingival graft; Procedure: Suture

INTERVENTIONS:
Procedure: Free gingival graft — 1.5-2 x 5 x 10 mm size epithelialized graft harvested from the palate is stabilized in the mandibular anterior single-tooth recession region
Procedure: Cyanoacrylate — N-Butyl-Cyanoacryle is applied to stabilize the graft to the recipient bed and to coat the donor site wound
  Arms: Cyanoacrylate
Procedure: Suture — The graft is stabilized with 6/0 polyvinylidene fluoride suture to the recipient bed
  Arms: Suture

SUMMARY:
Present study aims to reveal the effects of cyanoacrylate application at the recipient bed and the donor site in free gingival graft surgery on the healing parameters and patient-based outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Single-tooth gingival recession in the anterior mandibular region
* Pain with chewing or oral hygiene practice
* Ongoing recession

Exclusion Criteria:

* Systemic disease
* Smoking
* Pregnancy / lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Re-epithelization | one week after the surgery
  Donor site re-epithelization: hydrogen-peroxide is applied to the donor area with the help of an injector, and it is recorded as complete when no foaming occurs
Re-epithelization | two weeks after the surgery
  Donor site re-epithelization: hydrogen-peroxide is applied to the donor area with the help of an injector, and it is recorded as complete when no foaming occurs
Re-epithelization | three weeks after the surgery
  Donor site re-epithelization: hydrogen-peroxide is applied to the donor area with the help of an injector, and it is recorded as complete when no foaming occurs
Post-operative pain | 1st week
  Visual analogue scale (VAS) (0-10), self-reported outcome 0 - no pain (min.) 10 - unbearable (max.)
Post-operative pain | 2nd week
  Visual analogue scale (VAS) (0-10), self-reported outcome 0 - no pain (min.) 10 - unbearable (max.)
Post-operative pain | 3rd week
  Visual analogue scale (VAS) (0-10), self-reported outcome 0 - no pain (min.) 10 - unbearable (max.)
Post-operative pain | 4th week
  Visual analogue scale (VAS) (0-10), self-reported outcome 0 - no pain (min.) 10 - unbearable (max.)
Oral health impact profile (OHIP-14) | Baseline
  The patients are asked to fill provided OHIP-14 forms Questionnaire about satisfaction related to oral health, scored as 0-4 (never - always) 14 questions in total 0 (min.) - 56 (max.) Lower scores represent higher oral health related life quality
Oral health impact profile (OHIP-14) | 3rd day
  The patients are asked to fill provided OHIP-14 forms Questionnaire about satisfaction related to oral health, scored as 0-4 (never - always) 14 questions in total 0 (min.) - 56 (max.) Lower scores represent higher oral health related life quality
Oral health impact profile (OHIP-14) | 1st week
  The patients are asked to fill provided OHIP-14 forms Questionnaire about satisfaction related to oral health, scored as 0-4 (never - always) 14 questions in total 0 (min.) - 56 (max.) Lower scores represent higher oral health related life quality
Oral health impact profile (OHIP-14) | 1st month
  The patients are asked to fill provided OHIP-14 forms Questionnaire about satisfaction related to oral health, scored as 0-4 (never - always) 14 questions in total 0 (min.) - 56 (max.) Lower scores represent higher oral health related life quality
Graft dimensions | 1st month
  Mesio-distal (horizontal) and apico-coronal (vertical) width of the graft is measured with a periodontal probe, rounding to the nearest mm
Graft dimensions | 3rd month
  Mesio-distal (horizontal) and apico-coronal (vertical) width of the graft is measured with a periodontal probe, rounding to the nearest mm
Graft dimensions | 6th month
  Mesio-distal (horizontal) and apico-coronal (vertical) width of the graft is measured with a periodontal probe, rounding to the nearest mm

SECONDARY OUTCOMES:
Mucosal thickness | In the beginning of the surgery (baseline)
  15 endodontic reamer is inserted to the palatal mucosa 5 mm apical of the gingival margin of the second premolar; under local anesthesia
Paresthesia / hyperesthesia in the donor site | 1st month
  The patient marks the visual analogue scale (0-10) after rubbing the donor site with a periodontal probe (to give a reference, symmetrical area is rubbed first) 0 - Paresthesia / hyperesthesia, 10 - no sensation difference with the reference area
Color harmony | 1st week
  Color harmony between the graft and the neighboring keratinized tissue at the recipient site, examiner gives a score ranging 0-10 0 - completely different tone/color of the graft; 10 - no detectible tone difference
Color harmony | 2nd week
  Color harmony between the graft and the neighboring keratinized tissue at the recipient site, examiner gives a score ranging 0-10 0 - completely different tone/color of the graft; 10 - no detectible tone difference
Color harmony | 1st month
  Color harmony between the graft and the neighboring keratinized tissue at the recipient site, examiner gives a score ranging 0-10 0 - completely different tone/color of the graft; 10 - no detectible tone difference
Color harmony | 3rd month
  Color harmony between the graft and the neighboring keratinized tissue at the recipient site, examiner gives a score ranging 0-10 0 - completely different tone/color of the graft; 10 - no detectible tone difference
Color harmony | 6th month
  Color harmony between the graft and the neighboring keratinized tissue at the recipient site, examiner gives a score ranging 0-10 0 - completely different tone/color of the graft; 10 - no detectible tone difference

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa YILMAZ, PhD, Principal Investigator — Biruni University, assistant professor
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared
Supporting Information: Study Protocol
Time Frame: one year after the publication